CLINICAL TRIAL: NCT00223028
Title: Investigation of the Steady State Pharmacokinetics of Sirolimus, Mycophenolat Mofetil and Fluvastatin After Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2004-07

CONDITIONS: Renal Transplantation
Keywords: fluvastain; sirolimus; mycophenolat mofetil; renal transplantation
MeSH Terms: interventions — Sirolimus; Fluvastatin

INTERVENTIONS:
Drug: sirolimus, mycophenolat mofetil, fluvastatin

SUMMARY:
To investigate in renal transplant recipients the potential drug intreaction between Sirolimus, Mycophenolt Mofetil and Fluvastatin

All patient enrolled in this PKI-Study had no changes in the therapy before or because of the study. Only patients without changes more than 4 weeks before startin the study were included

ELIGIBILITY:
Inclusion Criteria:

* renal transplant patients (18 - 65 years, inclusive)
* cadaver and living renal transplants(1. Ntx, 2. Ntx)
* Immunsuppression: sirolimus with or without Mycophenolat Mofetil und and fluvastatin Fluvastatin for a minimum of three months
* writen informt consent by the patient

Exclusion Criteria:

* contraindications for statins
* pregnancy or lactating
* elevated liver or muscle encymes (> 2x up to normal values: AST, ALT, bilirubine, CPK)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-04; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Renders, MD, Principal Investigator — University of Schleswig-Holstein, Campus Kiel, Department of Nephrology